CLINICAL TRIAL: NCT00873509
Title: A Randomized, Placebo-controlled, Double-masked Clinical Trial of Buspirone in the Treatment of 2- 6 Year Old Children With Autistic Disorder
Brief Title: Buspirone in the Treatment of 2-6 Year Old Children With Autistic Disorder
Acronym: B-ACE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chugani, Diane C. (Individual)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Diane C Chugani, Chief, Division of Clinical Pharmacology and Toxicology, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10888; 5U01NS061264 (NIH)
Record Dates: First submitted 2009-03-30; First posted 2009-04-01 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Autistic Disorder
Keywords: Autism
MeSH Terms: conditions — Autistic Disorder | interventions — Buspirone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Buspirone 2.5 mg
  Interventions: Drug: Buspirone
- 2 (Experimental): Buspirone 5.0 mg
  Interventions: Drug: Buspirone
- 3 (Placebo Comparator): Placebo match
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Buspirone — Buspirone liquid, 2.5 mg in 1 ml, once per day in the evening for the first week of administration and thereafter twice a day 12 hours apart for the entire study
  Arms: 1
Drug: Buspirone — Buspirone liquid, 5.0 mg in 1 ml , once per day in the evening for the first week of administration and thereafter twice a day 12 hours apart for the entire study
  Arms: 2
Drug: Placebo — Placebo liquid, in 1 ml, once per day in the evening for the first week of administration and thereafter twice a day 12 hours apart for the entire study
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate the effects of twice-daily oral buspirone on core features of autism in autistic children aged 2-6 years as measured by the change from baseline in the Autism Diagnostic Observation Schedule (ADOS) Composite Total scores compared to placebo at 6 months.

DETAILED DESCRIPTION:
This is a multi-center, randomized, placebo-controlled, double-masked study of 166 evaluable participants taking buspirone twice daily for 6 months. Children aged 2-6 years with autism will be randomized to receive one of three treatments: 2.5mg, 5.0mg, or matched placebo. The placebo controlled trial will be followed by an optional follow-up trial to assess the long term safety of buspirone. In addition, a PET scan of serotonin synthesis and plasma serotonin will be measured at baseline to determine whether these measures are predictors of drug response. This trial is aimed at the core features of autism. The outcome measures for efficacy will be examiner and parent ratings on psychological tests and questionnaires. The outcome measure for the primary objective will be the Autism Diagnostic Observation Scale (ADOS) Composite Total score. The behavioral outcomes for the secondary aims are delineated in the study design.

ELIGIBILITY:
Inclusion Criteria:

* Participants: must meet the study definition for diagnosis of autistic disorder as determined by clinical diagnosis based upon DSM-IV criteria, the Autism Diagnostic Interview-Revised (ADI-R) and the Autism Diagnostic Observation Schedule (ADOS) performed at baseline 1. ADI-R will be conducted by trained study staff at Baseline 1 Visit. If the participant has had an ADI-R in the past 12 months, this will be accepted provided the person administering and scoring the test is site personnel validated for the study.
* Age 2 to less than 6 years, male and female.
* Parent/Legal Guardian/Caregiver must be able to understand , read and speak English
* Written Informed Consent.

Exclusion Criteria:

* Presence or history of neurological disorders, including seizure disorders (abnormal EEG without seizures will not be excluded), PKU, tuberous sclerosis, Rett syndrome, Fragile X syndrome, Down Syndrome and traumatic brain injury.
* Other medical or behavioral problems requiring medications which are centrally active.
* Clinical or laboratory evidence of renal or hepatic disease (SGPT, GGT > 2 x normal value, and serum creatinine > 1.5 x normal value).

Treatment with any medication known to alter the activity of the CYP3A4 enzyme including ketoconazole, itraconazole, grapefruit juice, erythromycin, clarithromycin, cimetidine, verapamil, diltiazem, rifampin, phenytoin, phenobarbital, or carbamazepine within the previous 2 months and for the duration of the study is prohibited.

* Use of centrally acting drugs during the 6 weeks prior or during the study. These drugs include but are not limited to neuroleptics, benzodiazepines, anticonvulsants and antidepressants. Shorter times may be considered depending on the half life of the drug.
* Prior treatment for periods longer than two weeks with buspirone or selective serotonin reuptake inhibitors. This includes herbal substances such as St John's Wort which have similar pharmacological actions.
* Known allergies to study medication.
* Unable to provide the required blood samples.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 166 (Actual)
Dates: Start 2009-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of twice-daily oral buspirone on core features of autism in autistic children 2-6 years measuring the change from baseline in ADOS (Autism Diagnostic Observation Schedule) Composite Total scores compared to placebo at 6 months. | Baseline 1, Week 24

SECONDARY OUTCOMES:
To evaluate the effects of twice-daily oral buspirone on the ADOS Composite calibrated severity score, social behavior, repetitive behavior, language, sensory dysfunction and anxiety. | Baseline 1, Week 24 and Week 48
To determine whether there are age group differences in the effects of buspirone on social interaction, repetitive behavior, language, sensory dysfunction and anxiety. | Baseline 1, Week 1, Week 24, Week 48
To determine whether there is a difference in the incidence of side effects and long term safety between the buspirone and placebo groups, and between the different dose groups. | Duration of the study
To determine whether the whole brain PET measure of serotonin synthesis capacity is a predictor of buspirone effect. | Baseline 2
To determine whether blood serotonin concentration is a predictor of buspirone effect. | Baseline 2

CONTACTS AND LOCATIONS:
Overall Officials: Diane C Chugani, PhD, Principal Investigator — Wayne State University
Locations (6):
- United States (6):
  - University California Davis M.I.N.D. Institute, Sacramento, California
  - Children's Hospital of Michigan Wayne State University, Detroit, Michigan
  - New York University Langone Medical Center, New York, New York
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic Lerner College of Medicine, Cleveland, Ohio
  - University of Texas Southwestern, Dallas, Texas

REFERENCES:
- [Result] Chugani DC, Chugani HT, Wiznitzer M, Parikh S, Evans PA, Hansen RL, Nass R, Janisse JJ, Dixon-Thomas P, Behen M, Rothermel R, Parker JS, Kumar A, Muzik O, Edwards DJ, Hirtz D; Autism Center of Excellence Network. Efficacy of Low-Dose Buspirone for Restricted and Repetitive Behavior in Young Children with Autism Spectrum Disorder: A Randomized Trial. J Pediatr. 2016 Mar;170:45-53.e1-4. doi: 10.1016/j.jpeds.2015.11.033. Epub 2015 Dec 30. PMID 26746121
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711
- Available data/document: Individual Participant Data Set — https://ndar.nih.gov